CLINICAL TRIAL: NCT03468192
Title: Hip Precautions Not Meaningful After Hemiarthroplasty Due to Hip Fracture. Cluster-randomized Study of 394 Patients Operated With Direct Anterolateral Approach.
Brief Title: Cluster-randomized Study of 394 Patients Operated With Direct Anterolateral Approach.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Ammar Jobory, MD, PhD student, Lund University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AmmarJobory
Record Dates: First submitted 2018-02-12; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Intervention Model Description: Cluster-randomized study of 394 patients operated with direct anterolateral approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-precaution group (Experimental): Study Group: Patients in the NPG had no restrictions on mobility, i.e. they were encouraged to move freely during the recovery phase and assistive equipment were prescribed only if needed.
  Interventions: Other: Non-precaution group
- precaution group (No Intervention): Control Group: the precaution group (PG) had standard postoperative hip precautions included limited flexion of the hip to 90° (avoid reaching down to toes or bringing knee up beyond 90°) and limited adduction of the hip (avoid sleeping on side and avoid crossing legs at knees or ankles). The mandatory assistive equipment to use for at least 3 months were reacher and stocking application aid. The patients were instructed only to use elevated chair, bed and toilet in order not to flex more than 90° in the hip. For the same reason a brace over the knee was prescribed for 6 weeks, particularly in patients with cognitive limitations.

INTERVENTIONS:
Other: Non-precaution group — Patients in the NPG had no restrictions on mobility, i.e. they were encouraged to move freely during the recovery phase and assistive equipment were prescribed only if needed
  Arms: non-precaution group

SUMMARY:
394 participants were cluster-randomized during 2010-2014. Depending on which ward the participants admitted to, they were allotted to free rehabilitation (non-precaution group, NPG, n=226) or our conventional regime with precautions and mandatory assistive equipment (precaution group, PG, n=168). The participants were followed during hospital stay, at 6 weeks (postal questionnaire), 3 month (visit) and 6 months (reading of medical records) by means of function tests, health-related quality of life (EQ-5D) and other patient-reported outcome measures (PROM).

DETAILED DESCRIPTION:
394 participants with Garden III-IV (20) femoral neck fractures treated with hemiarthroplasty participated in a cluster-randomised study during 2010-2014 at Skane University Hospital, Malmö. Inclusion criteria was an acute displaced femoral neck fracture treated with a bipolar hemiarthroplasty inserted via a direct lateral approach in supine position. All such participants were considered potential study participants and invited to the study by an occupational therapist (OT), within the first postoperative days. If the participants was not capable of making decisions, relatives were asked. The study was approved by The Regional Ethical Review Board in Lund on condition that all participants, regardless of group, or their next-in-kin gave written consent (Dnr 2009/754).

The four wards managing hip fracture patients were assigned either to provide the standard postoperative hip precaution regime or the non-precaution regime during the entire study period. In two of the wards, the precaution group (PG) had standard postoperative hip precautions included limited flexion of the hip to 90° (avoid reaching down to toes or bringing knee up beyond 90°) and limited adduction of the hip (avoid sleeping on side and avoid crossing legs at knees or ankles). The mandatory assistive equipment to use for at least 3 months were reacher and stocking application aid. The participants were instructed only to use elevated chair, bed and toilet in order not to flex more than 90° in the hip. For the same reason a brace over the knee was prescribed for 6 weeks, particularly in participants with cognitive limitations.

The non-precaution group (NPG) consisted of participants treated in the other two wards. Participants in the NPG had no restrictions on mobility, i.e. they were encouraged to move freely during the recovery phase and assistive equipment were prescribed only if needed.

Admittance of a participant to either ward was only decided by any available bed, i.e. the health status of the participants or any other factors did not influence placement of participants. The investigators recruited 168 participants to the PG and 226 participants to the NPG.

The initial power analysis was directed towards dislocation rate as primary outcome. When designing the trial, the investigators had a dislocation rate of 0.5% at the department. The investigators calculated that, in order to detect an increase of 3.5%, i.e. a clinical relevant effect, the investigators needed 340 participants in each group (p<0.05). The original plan was to additionally monitor PROM in the first 400 participants, and then dislocation rate only in the remaining 400. In order to monitor the safety of the study, the investigators also calculated a non-inferiority model, with warning levels at which the investigatorswould discontinue the study. This model was based on 200 participants in each group. Due to recruitment difficulties, the study was closed after inclusion of approximately 400 participants.

Both groups had functional assessment by an OT done as part of standard-of-care, usually within the three first postoperative days. The surgical procedure was a bipolar hemiarthroplasty inserted via a direct lateral approach (Hardinge). All implants were cemented, except 5 in the NPG and 2 in the PG (2.2 and 1.2 %).

During hospital stay the investigators registered time from admission to surgery, time of surgery, type of implant, adversities during surgery, the experience of the surgeon, radiological evaluation, length of stay, any deaths and dismissal address. The work burden of the rehabilitation personnel during hospital stay was estimated by themselves as "very short", "short", "normal", "long" or "very long" work effort. No one reported "very long". "Very short" and "short" was grouped together in the analyses. The participants were followed up with postal questionnaire at 6 weeks and 3 months including EQ-5D and a visual analogue scale on pain and satisfaction (0 to 100). A physiotherapist assessed participants with functional tests at 3 months. As only half of participants chose to participate in functional testing, the investigators do not report these data.

Medical records from all somatic departments of the hospital were reviewed and all adverse events (death, dislocation, surgical site infection (SSI), periprosthetic fracture, deep vein thrombosis, pulmonary embolism, pneumonia, falls and new fractures, stroke and ischemic heart attack) up to 6 months postoperatively were recorded. SSI was divided in to superficial incisional SSI and deep incisional SSI and were defined according to Horan et al.The follow-up cannot consider to be blinded, as some results were gathered during hospital stay were the group belonging of the participants were obvious.

ELIGIBILITY:
Inclusion Criteria:

* patients with Garden III-IV (20) femoral neck fractures treated with hemiarthroplasty participated in a cluster-randomised study during 2010-2014.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Dislocation | 6 months
  Dislocation of prosthesis identifed on x-ray

SECONDARY OUTCOMES:
PROM | 3 months
  EQ5D

IPD SHARING:
Plan to Share IPD: Undecided